CLINICAL TRIAL: NCT01717443
Title: The Incidence, Prevalence and Genotype of Genital Human Papillomavirus Infections in Females Before and After Renal Transplantation
Brief Title: Genital HPV Infections Before and After Renal Transplantation
Status: Completed | Type: Observational
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Principal Investigator, Joanne A. de Hullu, MD, PhD, MD, PhD, University Medical Center Nijmegen
Other Study IDs: NL38266.091.11
Record Dates: First submitted 2012-08-23; First posted 2012-10-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Human Papillomavirus Infections
Keywords: Human Papillomavirus; Renal transplantation
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women, renal disease, transplantation: Women with end-stage renal disease, whose eligibility for renal transplantation is assessed

SUMMARY:
The purpose of this study is to examine the prevalence, incidence and genotype of anogenital HPV infections in women before and after renal transplantation. With this information the investigators can determine the value of vaccination in patients waiting for renal transplantation in the future.

DETAILED DESCRIPTION:
Each year about 800 renal transplantations are performed in the Netherlands. The current immunosuppressive strategies have led to a 1-year patient and graft survival of more than 90%. This high survival rate urges medical specialists to pay increasing attention to the long-term side effects of immunosuppressive medication, such as virus-associated cancers. An example of an oncogenic virus is the high risk Human Papillomavirus (hrHPV) which is related to (pre)malignancies of the anogenital tract e.g. cervix, vulva and anus. These malignancies are among the most common malignancies in renal transplant recipients (RTRs). The incidence of hrHPV-related cervical and vulvar malignancies is increased up to a 100-fold in RTRs compared to the general population. There is limited literature on the exact behaviour of HPV infection related anogenital (pre)malignancies in RTRs. A part of these (pre)malignancies are probably already present at the time of transplantation while others develop in the years after transplantation. With gynaecological examination the investigators can diagnose anogenital (pre)malignancies before transplantation so treatment, if necessary, can commence before transplantation. Knowledge about HPV status before and after transplantation gives insight in the natural course of the HPV infection in this group of patients and with this information the investigators can determine the value of vaccination in patients waiting for renal transplantation in the future.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Age ≥ 18 years at start of the study;
* Eligible for renal transplantation;
* Operation at the Radboud University Nijmegen Medical Centre;
* Signed informed consent;
* Mentally capable to understand and comprehend the study and its implications;
* Sufficient knowledge of the Dutch language to read, fully understand and complete the Questionnaire.

Exclusion Criteria:

* Patient not willing to sign and/or return the informed consent form;
* Patient refusing additional treatment in case of abnormal findings at the first visit;
* Patient being pregnant, or within a period of 3 months after delivery;
* Patient being within a period of 3 months after miscarriage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of women above 18 years of age with end stage renal disease who are registered for renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of genital HPV infection before and after renal transplantation in women with end stage renal disease | 6 months before and 6 months after renal transplantation
  The difference between post-transplantation prevalence (two HPV tests in 6 months after transplantation)and pre-transplantation prevalence (two HPV tests in 6 months before transplantation) will be compared.

SECONDARY OUTCOMES:
Incidence of genital HPV infection before and after renal transplantation | Assessed every 3 months for 2 years
Genotype of the HPV infection per time point | Assessed every 3 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joanne A de Hullu, MD, PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands